CLINICAL TRIAL: NCT05684575
Title: Early Return of COVID-19 Patients to Home on Oxygen: Evaluation of a New Strategy Based on the City/hospital Link
Brief Title: Evaluation of the Outcome of COVID-19 Patients Discharged Home on Oxygen Therapy
Acronym: COVAMBU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRD1921
Record Dates: First submitted 2023-01-12; First posted 2023-01-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: COVID-19; Oxygen therapy; Early return
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phone satisfaction questionnaire (Other): Evaluation of the outcome of Covid-19 patients discharged home on oxygen therapy
  Interventions: Other: Phone satisfaction questionnaire

INTERVENTIONS:
Other: Phone satisfaction questionnaire — Evaluation of the outcome of Covid-19 patients discharged home on oxygen therapy

SUMMARY:
The René Dubos Hospital in Pontoise has set up a home discharge system for oxygen-requiring patients in collaboration with PRADO, a health insurance organization, or private providers. This organization coordinates the care to be implemented at home based on the city/hospital link. The coordinator of this organization was also in charge of scheduling a follow-up consultation between 7 and 14 days after hospital discharge.

The aim of this study is to evaluate this new organization, both in terms of its impact on patient outcomes (survival and re-hospitalization rates) and on patients' experiences and satisfaction with their care.

DETAILED DESCRIPTION:
The COVID-19 pandemic was responsible for an unprecedented hospital tension with multiple consequences (medical, economic, social...). The first scientific responses were found with unprecedented speed. Very quickly, innovative solutions and a complete reorganization of the health system were necessary to manage this crisis. In order to limit the number of patients hospitalized and/or the length of their hospitalization, most hospitals quickly set up systems to organize the early return of patients to their homes on oxygen. Studies evaluating telemedicine as a tool for monitoring oxygen-requiring patients at home have shown that it is effective and safe for monitoring these patients. Another retrospective study estimated the 30-day rehospitalization rate for patients with SARS-CoV-2 pneumonia after return home on oxygen with telephone monitoring by a nurse to be 8.5% (95% confidence interval, 6.2%-10.7%) and all-cause mortality to be 1.3% (95% confidence interval, 0.6%-2.5%).

The René Dubos Hospital in Pontoise has set up a home discharge system for oxygen-requiring patients in collaboration with PRADO, a health insurance organization, and a private provider. These organizations coordinate the care to be implemented at home based on the city/hospital link (oxygen provider, private nurse for the injection of anticoagulants and sometimes insulin and monitoring of vital parameters). These organizations were also in charge of scheduling a follow-up consultation between 7 and 14 days after hospital discharge, with the attending physician or, failing that, in the infectious diseases department of the Pontoise Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age

  * Patients with virologically proven COVID 19 (positive Polymerase Chain Reaction or antigenic test) or based on clinical and radiological evidence
  * Patients discharged from hospital or from the emergency room on oxygen between 1 and 5L at the time of discharge
  * Organization of discharge by a service provider (PRADO or private)

Exclusion Criteria:

* Patients discharged from the intensive care unit
* Oxygen-requiring patients > 5 Liters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Description of the evolution of patients with COVID-19 who benefited from an early return home on oxygen organized by the PRADO or a private provider | At 30 days of hospital discharge (D30)
  Assessment of mortality (all causes) at 30 days of hospital discharge (D30) : number of died patients

SECONDARY OUTCOMES:
Assessment of the risk of early re-hospitalization of patients following their return home | At 7 days from hospital discharge (D7)
  Number of re-hospitalizations at 7 days from hospital discharge (D7)
Assessment of patients' satisfaction with their care and return home | At the end of the study, an average of 10 month
  Evaluation of patients'satisfaction :
  Satisfaction questionnaire contains 5 questions :
  For Q1, patient answer : Very satisfied, Satisfied, Neither satisfied or unsatisfied, Unsatisfied or Very unsatisfied For Q2, patient answer : Very confident, Confident, Neither confident or anguished, Anguished or Very anguished For Q3, patient answer : Yes, I don't know or No For Q4 and Q5, patient answer : Yes or No

CONTACTS AND LOCATIONS:
Overall Officials: Dr Celeste Lambert, Principal Investigator — Hospital René Dubos Pontoise
Locations (2):
- France (2):
  - Polyvalent, infectious and pulmonary medicine - GHCPO Beaumont/Oise, Beaumont-sur-Oise
  - Aval-emergency medicine department - Infectious diseases departement- Hospital René Dubos Pontoise, Pontoise

IPD SHARING:
Plan to Share IPD: No